CLINICAL TRIAL: NCT05656014
Title: The Relationship of Medial Longitudinal Arch Height With Pain, Disease Severity and Knee Joint Alignment in Patients With Knee Osteoarthritis
Brief Title: The Relationship of the Medial Longitudinal Arch Height With Clinical Features of Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Levent Karataş, Investigator, MD, Gazi University
Other Study IDs: Knee osteoarthritis and AHI
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Foot Deformities; Pes Planus; Pes Cavus; Knee Osteoarthritis; Knee Pain Chronic; Disability Physical; Lower Limb Deformity
Keywords: Medial longitudinal arch; Arch height index; Knee osteoarthritis; Knee pain; Foot; Lower limb alignment
MeSH Terms: conditions — Foot Deformities; Flatfoot; Talipes Cavus; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with knee osteoarthritis: Adult patients 50 years of age or older diagnosed with knee osteoarthritis according to American College of Rheumatology criteria

SUMMARY:
The goal of this observational study is to investigate the relationships between the medial longitudinal arch (MLA) height of the foot and clinical and radiological characteristics of knee osteoarthritis in adult patients 50 aged and over. The main questions it aims to answer are:

* Is there any relationship between knee pain and disability in knee osteoarthritis and MLA height?
* Is there any relationship between the radiologic severity of knee osteoarthritis and MLA height?
* Is there any relationship between knee joint alignment in knee osteoarthritis and MLA height?

DETAILED DESCRIPTION:
Differences in hind and midfoot structures, including the medial longitudinal arch, affect lower limb alignment and biomechanics. However, the causal relationship between knee joint problems and foot deformities is controversial. Knee osteoarthritis, a common orthopaedic condition in the elderly population, tends to distort the lower limb alignment by narrowing the tibiofemoral joint space asymmetrically. Therefore, knee varus and medial longitudinal arch deformities may change gait biomechanics on knee osteoarthritis. However, there is insufficient evidence on the relationship between variation in foot posture and disease severity, knee varus deformity, knee pain and disability in knee osteoarthritis. In this study, investigators will examine the lower extremity alignment and osteoarthritis severity in terms of MLA height in adults with knee osteoarthritis.

The study sample will be formed by the simple random sampling method from adult patients with knee osteoarthritis who will be admitted to our clinics and outpatient clinics with knee pain. It was planned to include 93 participants to be able to detect the two-way correlation between the knee WOMAC score and the arch height index with an effect size of 0.3, a power of 90%, and a 5% margin of error.

Initially, demographic data, including age, gender, body mass index (BMI), limb dominance, and time from knee pain onset of participants, will be recorded. For both knees goniometric measurement of knee passive range of motion (ROM), visual analogue scale (VAS) for pain and Western Ontario and McMaster Universities Arthritis Index (WOMAC) will be applied. Kellgren/Lawrence stages, mechanical, and anatomical tibiofemoral angles for knee joints will be obtained from lower limb length X-ray. MLA height index measurement will be performed by an investigator blinded to the patient's clinical condition. According to the results of descriptive statistics, the relationship between MLA height measurement results (arch height index and arch height flexibility) and Kellgren-Lawrence stage, VAS, WOMAC and tibiofemoral angles will be examined by correlation analysis. In case of significant correlation, regression analyses for Kellgren-Lawrence, VAS and WOMAC scores as dependent variables will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Being 50 years old or older
* Having a diagnosis of knee osteoarthritis according to the American College of Rheumatology

Exclusion Criteria:

* History of fracture or orthopaedic surgery involving lower limbs
* Presence of neurological condition resulting in lower limb sensorimotor deficit
* Having another inflammatory rheumatological disease
* Having a malignant tumour with bone metastasis
* Having lower limb oedema, lymphedema, skin and soft tissue loss that will prevent the evaluation of foot morphology (arch height index)
* Severe neuropsychiatric disease or condition that interferes with communication
* Having therapeutic injection into the knee joint in the last 3 months
* Presence of any major trauma that aggravated knee pain in the last 6 weeks

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 50 years of age or older diagnosed with osteoarthritis of one or both knees according to the American College of Rheumatology criteria
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Arch Height Index while bipedal standing | Within the three days of clinical evaluation
  The ratio of the dorsum height of the foot (measured in the middle of the total foot length) to truncated foot length, while bipedal standing. Normal values have been reported to be approximately 0.338 ± 0.031 to 0.343 ± 0.033 in college-aged women. Higher values represent the increased medial longitudinal arch height of the foot (e.g. pes cavus) while lower values are related to pes planus.
Arch Height Index while sitting | Within the three days of clinical evaluation
  The ratio of the dorsum height of the foot (measured in the middle of the total foot length) to truncated foot length, while sitting with feet calmly on the ground. Normal values have been reported to be approximately 0.355 ± 0.031 to 0.369 ± 0.034 in college-aged women. Higher values represent the increased medial longitudinal arch height of the foot (e.g. pes cavus) while lower values are related to pes planus.
Arch Height Flexibility | Within the three days of clinical evaluation
  Arch Height Flexibility will be calculated by the [(arch height while sitting - arch height while standing) / 0.4 x body weight] x 100 (m/kN) formula. Higher values represent the more flexible medial longitudinal arch structure.
Kellgren Lawrence stage of knee osteoarthritis | Within the three days of clinical evaluation
  It is a radiological grading of knee osteoarthritis with a value between 0 to 4. Medial and lateral tibiofemoral compartments are evaluated on weight-bearing anteroposterior knee radiograph in terms of joint space narrowing, subchondral periosteal sclerosis, subchondral cyst and osteophytic formations. Zero means no radiographic evidence of osteoarthritis, while 4 indicates advanced knee osteoarthritis.
Anatomical tibiofemoral angle | Within the three days of clinical evaluation
  It is the angle, measured on a weight-bearing, full-length anteroposterior lower limb radiograph, between the anatomical axes of the femur and tibia. The normal value of the anatomical tibiofemoral angle is between 4 to 6 degrees of valgus. A higher positive value will indicate more valgus posture of the knee, while lower or negative values will be related to varus deformity.
Mechanical tibiofemoral angle | Within the three days of clinical evaluation
  It is the angle, measured on a weight-bearing, full-length anteroposterior lower limb radiograph, between the lines drawn from the femoral head to the femoral intercondylar notch and from the tibial interspinous point to the tibial mid-plafond. The mechanical tibiofemoral angle is approximately 1-1.5 degrees of varus for a knee in normal alignment. In this study, to ensure consistency with the anatomical tibiofemoral angle values, the direction of angulation will be noted as a positive or negative value for the valgus or varus, respectively.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores for both knees | Within the three days of clinical evaluation
  WOMAC is a specific, valid and reliable tool for measuring disability in the knee and hip osteoarthritis. It includes 24 questions under three sub-domains: pain, stiffness, and physical function. Each question is scored on a Likert scale as 0=none, 1=mild, 2=moderate, 3=severe, and 4=extreme. The total score is defined by the [(sum of the scores)/96]x100 formula and ranges from 0 to 100. Higher scores indicate increased disability due to more severe pain, stiffness and impaired physical function.
Visual analogous scale score for knee pain | Within the three days of clinical evaluation
  Participants are asked to mark the severity of their right and left knee pain in the past month on a 100 mm horizontal line; where point zero represents "no pain" and point 100 represents "the most severe pain possible". The result is noted in millimetres by measuring the distance from the "zero" to the marked point. Increasing values represent higher pain intensity.

SECONDARY OUTCOMES:
Knee range of motions | Within the day of clinical evaluation
  Flexion and extension range of motions will be measured using a goniometer regarding the neutral zero method for both knees. Decreased values represent a limited range of motion of the knee joint.
Time after pain onset (weeks) | Within the day of clinical evaluation
  The duration of knee pain leading to hospital admission will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Karataş, MD, Principal Investigator — Gazi University Faculty of Medicine
Locations (1):
- Gazi University Hospital, Department of Physical Medicine and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Williams DS, McClay IS. Measurements used to characterize the foot and the medial longitudinal arch: reliability and validity. Phys Ther. 2000 Sep;80(9):864-71. PMID 10960934
- [Background] Weimar WH, Shroyer JF. Arch height index normative values of college-aged women using the arch height index measurement system. J Am Podiatr Med Assoc. 2013 May-Jun;103(3):213-7. doi: 10.7547/1030213. PMID 23697727
- [Background] Hillstrom HJ, Song J, Kraszewski AP, Hafer JF, Mootanah R, Dufour AB, Chow BS, Deland JT 3rd. Foot type biomechanics part 1: structure and function of the asymptomatic foot. Gait Posture. 2013 Mar;37(3):445-51. doi: 10.1016/j.gaitpost.2012.09.007. Epub 2012 Oct 26. PMID 23107625
- [Background] Zifchock RA, Theriot C, Hillstrom HJ, Song J, Neary M. The Relationship Between Arch Height and Arch FlexibilityA Proposed Arch Flexibility Classification System for the Description of Multidimensional Foot Structure. J Am Podiatr Med Assoc. 2017 Mar;107(2):119-123. doi: 10.7547/15-051. Epub 2017 Feb 15. PMID 28198638
- [Background] Karatas L, Vuralli D, Gunendi Z. The effect of medial longitudinal arch height and medial longitudinal arch support insoles on postural balance in perimenopausal women. Turk J Med Sci. 2019 Jun 18;49(3):755-760. doi: 10.3906/sag-1808-39. PMID 31023006
- [Background] Marques Luis N, Varatojo R. Radiological assessment of lower limb alignment. EFORT Open Rev. 2021 Jun 28;6(6):487-494. doi: 10.1302/2058-5241.6.210015. eCollection 2021 Jun. PMID 34267938
- [Background] Moreland JR, Bassett LW, Hanker GJ. Radiographic analysis of the axial alignment of the lower extremity. J Bone Joint Surg Am. 1987 Jun;69(5):745-9. PMID 3597474